CLINICAL TRIAL: NCT06621667
Title: Response of Lung Function, Chest Mobility, and Kyphotic Curve to Diaphragmatic Myofascial Release in Hyperkyphotic Subjects: A Randomized Controlled Trial
Brief Title: Diaphragmatic Myofascial Release for Hyperkyphotic Subjects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Shafiek Mustafa Saleh, assistance professor doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: myorelease for hyperkyphosis
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Hyperkyphosis
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental)
  Interventions: Other: diaphragmatic myofascial release with traditional physical therapy exercises for hyperkyphosis
- control group (Active Comparator)
  Interventions: Other: traditional physical therapy exercises for hyperkyphosis

INTERVENTIONS:
Other: diaphragmatic myofascial release with traditional physical therapy exercises for hyperkyphosis — diaphragmatic myofascial release
  Arms: study group
Other: traditional physical therapy exercises for hyperkyphosis — traditional physical therapy exercises for hyperkyphosis
  Arms: control group

SUMMARY:
kyphotic subjects have respiratory disturbances due to weakening of the diaphragm, responsible for inhalation, which lead to abnormalities in respiratory mechanics and abnormal gas exchange, leading to respiratory complications. Myofascial release of the diaphragm is an intervention intended to indirectly stretch the diaphragm muscle fibers to reduce muscle tension, normalize fiber length, and promote the efficiency of muscle contraction. Although diaphragm myofascial release has been used in clinical practice, to the best of the authors' knowledge, the current study is the first research investigating the effect of diaphragmatic myofascial release on lung function, chest mobility and kyphotic curve in hyperkyphotic subjects.

ELIGIBILITY:
Inclusion Criteria:

* The participant's age ranged from 20 to 40 years.
* kyphosis angle 40-50◦
* reporting pain on palpation of the diaphragm

Exclusion Criteria:

* A history of respiratory diseases, heart disease, vascular disease, central nervous system disorder, psychiatric disorders, hypertension.
* History of any trauma or fracture to the thoracic spine.
* inflammatory diseases such as rheumatoid arthritis, musculoskeletal problem and neurological deficit
* Restrictive respiratory disease, smokers.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
maximum voluntary ventilation | change from base line at 4 weeks.
  the maximum voluntary ventilation will be measured using spirometer

SECONDARY OUTCOMES:
Chest expansion | change from base line at 4 weeks.
  the chest expansion will be measured using tap measurement
kyphotic angle | change from base line at 4 weeks.
  the kyphotic angle will be measured with flexicurve